CLINICAL TRIAL: NCT00836563
Title: The Natural History of Upper Arm Vessels Following Forearm Loop Arteriovenous
Brief Title: Vascular Changes Following Forearm Loop Arteriovenous Graft Placement
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0444-08-EP
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Chronic Kidney Disease
Keywords: Hemodialysis; Arteriovenous Graft
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Forearm Arteriovenous Loop Graft: Participants with planned forearm loop arteriovenous graft placement for hemodialysis or forearm loop arteriovenous graft placed within the previous 7 days will have the upper arm vessels assessed following forearm loop arteriovenous graft placement for size changes and timing of changes.

SUMMARY:
This study will determine whether upper arm vessels increase in size following forearm loop arteriovenous graft placement and the timing of these changes.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether upper arm vessels increase in size following forearm loop arteriovenous graft placement, and if they do, characterize the timing of these changes.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 19 years
2. Planned forearm loop arteriovenous graft placement for hemodialysis or forearm loop arteriovenous graft placed within the previous 7 days.
3. Cephalic and/or basilic vein diameter greater than or equal to 2.5 mm at the antecubital fossa to the axilla prior to AVG placement

Exclusion Criteria:

1. Age less than 19 years
2. Hemodialysis access other than forearm loop graft surgery placement
3. Cephalic and/or basilic vein diameter less than 2.5 mm at any point from the antecubital fossa to the axilla
4. Prior hemodialysis access surgery in the arm receiving the forearm loop graft

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing forearm arteriovenous loop graft placement
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-01-10 (Actual); Primary Completion 2011-12-13 (Actual); Study Completion 2011-12-13 (Actual)

PRIMARY OUTCOMES:
Upper arm vein diameter | Six months
  50% increase in upper arm vein diameter

CONTACTS AND LOCATIONS:
Overall Officials: Troy J Plumb, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center/The Nebraska Medical Center, Omaha, Nebraska, United States